CLINICAL TRIAL: NCT04016571
Title: Parameters to Assess Response to Intra-Venous Antibiotic Treatment for Pulmonary Exacerbations in Cystic Fibrosis
Acronym: PRIVATE
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 210802
Record Dates: First submitted 2019-01-18; First posted 2019-07-11 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pulmonary Exacerbation; Antibiotics; Outcome measures
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Expectorated sputum and blood samples will be collected. Samples will be processed within 24 hours or stored at - 80°. Processing will remove any human DNA or HTA relevant material.
  Samples from participants who have given consent for samples to be for future research will be stored at - 80°C, in a locked freezer in a lab with keypad access. Access to the samples will be limited to researchers involved in the study. Standard University custodial arrangements will apply.
  For samples from individuals who did not give consent for samples to be stored for the purposes of future research, they will be disposed in accordance with the HTA's code of practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Cystic Fibrosis: All Adults with a confirmed diagnosis of Cystic Fibrosis being admitted for Intra-Venous Antibiotic Treatment of a Pulmonary Exacerbation
  This study is observational so no intervention will be carried out.

SUMMARY:
Cystic fibrosis (CF) is a multisystem disease characterized by viscid secretions in multiple organ systems. Lung infection and damage account for most of the disease burden. Acute changes in respiratory signs and symptoms termed Pulmonary Exacerbations require treatment with intravenous antibiotics and hospital admission. These episodes cause substantial disruption to people's lives and impact on lung function, quality of life and lifespan. Current treatment regimes require improvement but further study is needed to identify who might benefit from a different approach.

This observational study aims to assess if multi-dimensional measurements taken during treatment correspond with later treatment response. This may allow us to personalise treatment more effectively in the future and to better understand how individuals respond to treatment.

DETAILED DESCRIPTION:
Pulmonary Exacerbations in CF require treatment with intravenous (IV) antibiotics and hospital admission for between 10-21 days. These episodes cause substantial disruption to people's lives and impact on lung function, quality of life and lifespan.Robust evidence to support current treatment approaches is lacking with awareness that current regimes could be optimised.

As yet there is no model for predicting how patients with CF will respond to IV antibiotic treatment- other than clinical judgement and lung function response.This is due to lack of robust measures to identify clinical response at the time of treatment and safely predict later clinical outcomes. The heterogeneity of the 21st Century CF population means a multi-dimensional composite measure is needed. This study has therefore been designed to provide an overall picture of people's response including clinical, biochemical and patient related outcome measures. Using multi-dimensional assessment we hope the measures assessed in this study will give a better picture of how people feel and how they respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients attending the adult service with a confirmed diagnosis of CF by sweat test or genotype
2. Able to provide written informed consent
3. Able to understand and comply with protocol requirements and instructions
4. Confirmed Pulmonary Exacerbation requiring treatment with intravenous antibiotics using defined criteria (Physician and patient agreed need for admission for intravenous antibiotic treatment)

Exclusion Criteria:

1. Previous recipient of a lung or other solid organ transplant
2. Inability to complete questionnaires
3. Current enrolment in other investigational medicinal product randomised trial
4. Admission for reasons other than pulmonary exacerbation of CF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a confirmed diagnosis of Cystic Fibrosis being admitted for treatment with intravenous antibiotics for a pulmonary exacerbation using defined criteria (Physician and patient agreed need for admission for intravenous antibiotic treatment)
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | Change in lung function between baseline and day 0, Day 5 and Day 14 of treatment
  Lung function Measure

SECONDARY OUTCOMES:
Treatment Failure defined by need for further IV antibiotic treatment within 30 days | Need for a further course of IV antibiotics within 30 days of treatment completion
  The number of participants requiring a further course of IV antibiotics within 30 days
Change in Respiratory Symptoms | Change between Day 0, day 5 and day 14 of treatment
  Change in Respiratory Symptoms assessed by CF-Respiratory Symptom Diary
Physical activity levels (step count, distance walked, Lightly active minutes, Moderate velocity physical activity (MVPA) and Exercise) | Change between Day 0, day 5 and day 14 of treatment
  Change in Physical Activity Levels measured by consumable wearable device
Sleep parameters measured by consumable wearable device | Change between Day 0, day 5 and day 14 of treatment
  Change in time in bed, time asleep and time awake/restless (mins)
Change in serum inflammatory marker (C-Reactive Protein) | Change between Day 0, day 5 and day 14 of treatment
  Change in serum inflammatory marker (CRP)
Change in sputum inflammatory markers | Change between Day 0, day 5 and day 14 of treatment
  Change in sputum (Interleukins, Tumour Necrosis Factor-Alpha, Calprotectin and Human Mobility Growth Box Protein -1) inflammatory markers (measured in pg/ml)
Change in microbiological growth measured by culture | Change between Day 0, day 5 and day 14 of treatment
  Change in microbiological growth measured by culture
Change in microbiological community composition measured by microbiota analysis | Change between Day 0, day 5 and day 14 of treatment
  Change in microbiological relative abundance, dominance, evenness, diversity and richness
Change in 24 hour sputum volume | Change between Day 0, day 5 and day 14 of treatment
  Change in 24 hour sputum volume (mls)
Time to next exacerbation | Time to next course of intravenous antibiotics within 12 month follow up period (study end)
  Time to next exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Damian Dr Downey, MBBS MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast Regional Adult CF Centre, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to maintain confidentiality

REFERENCES:
- [Background] Heltshe SL, Goss CH, Thompson V, Sagel SD, Sanders DB, Marshall BC, Flume PA. Short-term and long-term response to pulmonary exacerbation treatment in cystic fibrosis. Thorax. 2016 Mar;71(3):223-9. doi: 10.1136/thoraxjnl-2014-206750. Epub 2015 Apr 24. PMID 25911223
- [Background] Britto MT, Kotagal UR, Hornung RW, Atherton HD, Tsevat J, Wilmott RW. Impact of recent pulmonary exacerbations on quality of life in patients with cystic fibrosis. Chest. 2002 Jan;121(1):64-72. doi: 10.1378/chest.121.1.64. PMID 11796433
- [Background] de Boer K, Vandemheen KL, Tullis E, Doucette S, Fergusson D, Freitag A, Paterson N, Jackson M, Lougheed MD, Kumar V, Aaron SD. Exacerbation frequency and clinical outcomes in adult patients with cystic fibrosis. Thorax. 2011 Aug;66(8):680-5. doi: 10.1136/thx.2011.161117. Epub 2011 Jun 15. PMID 21680566
- [Background] VanDevanter DR, Pasta DJ, Konstan MW. Treatment and demographic factors affecting time to next pulmonary exacerbation in cystic fibrosis. J Cyst Fibros. 2015 Nov;14(6):763-9. doi: 10.1016/j.jcf.2015.02.007. Epub 2015 Mar 6. PMID 25754096
- [Background] Sanders DB, Bittner RC, Rosenfeld M, Hoffman LR, Redding GJ, Goss CH. Failure to recover to baseline pulmonary function after cystic fibrosis pulmonary exacerbation. Am J Respir Crit Care Med. 2010 Sep 1;182(5):627-32. doi: 10.1164/rccm.200909-1421OC. Epub 2010 May 12. PMID 20463179
- [Background] Flume PA, Mogayzel PJ Jr, Robinson KA, Goss CH, Rosenblatt RL, Kuhn RJ, Marshall BC; Clinical Practice Guidelines for Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: treatment of pulmonary exacerbations. Am J Respir Crit Care Med. 2009 Nov 1;180(9):802-8. doi: 10.1164/rccm.200812-1845PP. Epub 2009 Sep 3. PMID 19729669
- [Background] VanDevanter DR, O'Riordan MA, Blumer JL, Konstan MW. Assessing time to pulmonary function benefit following antibiotic treatment of acute cystic fibrosis exacerbations. Respir Res. 2010 Oct 6;11(1):137. doi: 10.1186/1465-9921-11-137. PMID 20925941
- [Background] Collaco JM, Green DM, Cutting GR, Naughton KM, Mogayzel PJ Jr. Location and duration of treatment of cystic fibrosis respiratory exacerbations do not affect outcomes. Am J Respir Crit Care Med. 2010 Nov 1;182(9):1137-43. doi: 10.1164/rccm.201001-0057OC. Epub 2010 Jun 25. PMID 20581166
- [Background] Smith DJ, Badrick AC, Zakrzewski M, Krause L, Bell SC, Anderson GJ, Reid DW. Pyrosequencing reveals transient cystic fibrosis lung microbiome changes with intravenous antibiotics. Eur Respir J. 2014 Oct;44(4):922-30. doi: 10.1183/09031936.00203013. Epub 2014 Jul 17. PMID 25034564
- [Background] Heltshe SL, Goss CH. Optimising treatment of CF pulmonary exacerbation: a tough nut to crack. Thorax. 2016 Feb;71(2):101-2. doi: 10.1136/thoraxjnl-2015-208057. No abstract available. PMID 26769012
- [Background] Shoki AH, Mayer-Hamblett N, Wilcox PG, Sin DD, Quon BS. Systematic review of blood biomarkers in cystic fibrosis pulmonary exacerbations. Chest. 2013 Nov;144(5):1659-1670. doi: 10.1378/chest.13-0693. PMID 23868694
- [Background] McCourt F, O'Neill B, Logan I, Abbott J, Plant B, McCrum-Gardner E, McKeown S, Stuart Elborn J, Bradley JM. Indicators of pulmonary exacerbation in cystic fibrosis: A Delphi survey of patients and health professionals. J Cyst Fibros. 2015 Jan;14(1):90-6. doi: 10.1016/j.jcf.2014.06.007. Epub 2014 Aug 12. PMID 25127921
- [Background] Goss CH, Edwards TC, Ramsey BW, Aitken ML, Patrick DL. Patient-reported respiratory symptoms in cystic fibrosis. J Cyst Fibros. 2009 Jul;8(4):245-52. doi: 10.1016/j.jcf.2009.04.003. Epub 2009 May 29. PMID 19481983